CLINICAL TRIAL: NCT00360451
Title: Preventing Depression in School Children
Brief Title: Effectiveness of School-Based Cognitive Behavioral Therapy in Preventing Depression in Young Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01 MH0522070; 5R01MH052270 (NIH); DSIR CT-P
Record Dates: First submitted 2006-08-02; First posted 2006-08-04 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2008-08

CONDITIONS: Depression; Anxiety
Keywords: Prevention; Child; Adolescent; Parent
MeSH Terms: conditions — Depression; Anxiety Disorders

ARMS (3):
- 1 (Experimental): Adolescent only Penn Resiliency Program
  Interventions: Behavioral: Adolescent only Penn Resiliency Program (Adolescent PRP)
- 2 (Experimental): Adolescent plus parent Penn Resiliency Program
  Interventions: Behavioral: Adolescent only Penn Resiliency Program (Adolescent PRP); Behavioral: Parent Penn Resiliency Program (Parent PRP)
- 3 (No Intervention): Control

INTERVENTIONS:
Behavioral: Adolescent only Penn Resiliency Program (Adolescent PRP) — In adolescent PRP, students learn both cognitive skills (recognizing the link between beliefs and emotions, challenging negative beliefs with evidence, making accurate attributions for events, and accurately assessing the ramifications of negative events) and behavioral problem-solving skills (decision making, assertiveness and negotiation, social skills, and relaxation).
  Arms: 1; 2
Behavioral: Parent Penn Resiliency Program (Parent PRP) — Parent PRP teaches parents to model and reinforce the skills taught in the adolescent program.
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of the Penn Resiliency Program, a school-based cognitive behavioral depression prevention program for young adolescents.

DETAILED DESCRIPTION:
Depression is a serious illness that affects a person's mood, thoughts, and physical well-being. Research suggests that approximately one in five children meets criteria for a major depressive episode by the end of high school. These children are at increased risk for a wide range of social, psychological, physical, and achievement-related problems. Thus, the potential benefits of effective and highly transportable depression prevention programs are enormous. The Penn Resiliency Program (PRP) is a school-based group intervention that teaches cognitive behavioral and social problem-solving skills to young adolescents. This study will examine the effectiveness of PRP in preventing symptoms of depression and anxiety among a group of young adolescents.

Participants in this open label study will be randomly assigned to one of three groups: adolescent only PRP, adolescent plus parent PRP, or no treatment control. In adolescent PRP, students will be taught cognitive and behavioral problem solving skills by school counselors and teachers. Parents in PRP will be taught to model and reinforce the skills taught in the adolescent program. Participants in the adolescent program will attend twelve 90-minute group sessions after school hours. Participants in the parent program will attend six 90-minute group sessions. Adolescent participants will attend booster sessions twice per year for 2 to 3 years after the initial treatment has ended. Parents will attend one booster session per year during the follow-up phase. Adolescents' depression and anxiety symptoms will be assessed through questionnaires at baseline, post-treatment, and 6-month intervals for 2 to 3 years following the intervention. Adolescents will also complete questionnaires about their coping behaviors, feelings of hopelessness, and several other outcomes related to depression and anxiety in adolescence. Data will be collected once per year from parents and teachers. Adolescent participants will also be assessed for depression and anxiety disorders each year the child is in the study.

ELIGIBILITY:
Inclusion Criteria:

* Student with above average levels of depression and anxiety symptoms (students with average or below average symptoms will be enrolled into the study space permitting)

Exclusion Criteria:

* Not a student in a participating school
* Not a student in grades six through eight

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2002-09; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Adolescents' depressive symptoms by self-report | Measured at baseline, post-treatment, and 6-month follow-ups
Adolescents' symptoms of anxiety by self-report | Measured at baseline, post-treatment, and 6-month follow-ups
Adolescents' symptoms of depression and anxiety, including clinical levels of symptoms, as assessed by diagnostic interview | Measured at baseline and 6, 18, and 30-month follow-ups

SECONDARY OUTCOMES:
Adolescents' externalizing symptoms by teacher report | Measured at baseline and 6, 18, and 30-month follow-ups
Adolescents' attributional style by self-report | Measured at baseline and 6, 18, and 30-month follow-ups
Parental depression by self-report | Measured at baseline and 6, 18, and 30-month follow-ups
Parental anxiety by self-report | Measured at baseline and 6, 18, and 30-month follow-ups
Parental attributional style by self-report | Measured at baseline and 6, 18, and 30-month follow-ups

CONTACTS AND LOCATIONS:
Overall Officials: Martin E.P. Seligman, PhD, Principal Investigator — Positive Psychology Center, University of Pennsylvania; Jane E. Gillham, PhD, Study Director — Swarthmore College & University of Pennsylvania; Karen J. Reivich, PhD, Study Director — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Gillham JE, Reivich KJ, Brunwasser SM, Freres DR, Chajon ND, Kash-Macdonald VM, Chaplin TM, Abenavoli RM, Matlin SL, Gallop RJ, Seligman ME. Evaluation of a group cognitive-behavioral depression prevention program for young adolescents: a randomized effectiveness trial. J Clin Child Adolesc Psychol. 2012;41(5):621-39. doi: 10.1080/15374416.2012.706517. Epub 2012 Aug 13. PMID 22889296